CLINICAL TRIAL: NCT06150404
Title: Parents' Voice and White Noises in Neonatal Intensive Care Unit: Efficacy Evaluation Against Noises' Damage - a Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial to Evaluate the Effect of White Noises and Parental Voices As Protectors Against Noise Damage in a Neonatal Intensive Care Unit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: From the preliminary data analysis, some unexpected results emerged that conducted us to terminate the enrollment.
Sponsor: Istituto Giannina Gaslini (Other)
Collaborators: Eubrain (Unknown)
Responsible Party: Principal Investigator, Silvia Rossi, Doctor in Methodology Research in Nursing, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SR-WHTNSS1
Record Dates: First submitted 2023-11-13; First posted 2023-11-29 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Premature Infant Disease
Keywords: premature; nursing care; randomized controlled trial; developmental care; noises damage; Newborn intensive care unit; white noises; parental voices
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Participation in intervention or control groups will occur using simple randomization techniques. Randomization will be achieved by creating a randomization list using specialized software. The randomization algorithm will be protected. The allocation sequence will be done using sealed opaque envelopes (making it impossible to read the contents), each numbered sequentially, containing the indication of assignment to the intervention group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Those in the intervention group will receive the administration of white noises and maternal and/or paternal voice recording.
  Interventions: Behavioral: White Noises and Maternal and/or Paternal voices
- Control Group (No Intervention): Those enrolled in the control group will receive standard care and will be subjected to the usual level of ambient noise.

INTERVENTIONS:
Behavioral: White Noises and Maternal and/or Paternal voices — The intervention group will receive white noise and maternal and/or paternal voice for a maximum of 4 hours per day, alternated as follows: 1 hour and 30 minutes of white noise, 30 minutes of maternal and/or paternal voice, 1-hour break, 1 hour and 30 minutes of white noise, 30 minutes of maternal and/or paternal voice. The intervention is expected to start at 08:00 in the morning and conclude at 13:00 and will be delivered from the day after the enrollment - when the parents provide their voice recording - until the day of discharge.
  The device for administering white noise and maternal and/or paternal voice will be placed approximately 30 cm from the head of the infant in the incubator and at the foot of the infant in the open crib.
  The volume will be 45 dB for infants in incubators and infants in open cribs.
  Arms: Intervention Group

SUMMARY:
The goal of this Randomized Controlled Trial is to test the efficacy of listening to white noises and parental voices against environmental noise damage in premature babies admitted to the Newborn Intensive Care Unit.

The main question it aims to answer is:

• Could the combined use of white noises and maternal and/or paternal voices reduce the negative outcomes of continuous exposure to hospital noises on newborns hospitalized in a Neonatal Intensive Care Unit?

Participants in the intervention group will listen to a recorded track composed of white noises and voices of their parents who read a story or sing a lullaby from the day of enrollment until the day of discharge, for 4 hours per day.

Researchers will compare the intervention group with the control group (who will receive the usual care provided without any intervention on the noise level) to see if babies enrolled in the intervention group show fewer events of tachycardia, tachypnea, desaturation, apnoea, and language or hearing impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the NICU with gestational age at birth ≥ 31 weeks (as this is the age at which sound perception is ≥ 40 dB and there is predictable clinical stability to allow intervention delivery without excessive interruptions)
* Patients admitted to the NICU who reach gestational age ≥ 31 weeks
* Patients monitored with the following types of monitors: Masimo rainbow SET™ (Masimo); Infinity® Delta (Draeger); Infinity® Acute Care System (Draeger); Efficia CM (Philips).

Exclusion Criteria:

* Patients with gestational age at birth < 31 weeks
* Patients affected by meningitis or severe cerebral insults, congenital brain anomalies, congenital syndromes with suspected or known brain dysfunction
* Patients diagnosed with hypoxic-ischemic encephalopathy
* Patients with significant airway abnormalities resulting in altered breathing during sleep
* Patients with terminal illnesses
* Patients with congenital anomalies of the face, ears, skull, or brain
* Patients with non-bacterial congenital infections
* Patients with congenital hearing deficits
* Patients whose parents or legal guardians refuse to participate in the study
* Patients already enrolled in other clinical studies.

Min Age: 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction of heart rate alteration | Through study completion, an average of 2 year
  Reduction, in the patients enrolled in the intervention group compared to the control group, in episodes of heart rate alteration associated with noises > 45 dB (nursing diagnosis: risk of tachycardia - HR >180 bpm - correlated with environmental exposure to noises > 45dB).
Reduction of oxygen saturation alteration | Through study completion, an average of 2 year
  Reduction, in the patients enrolled in the intervention group compared to the control group, in episodes of oxygen saturation alteration associated with noises > 45 dB (nursing diagnosis: risk of desaturation - SpO2 <90% - correlated with environmental exposure to noises > 45dB).
Reduction of respiratory rate alteration | Through study completion, an average of 2 year
  Reduction, in the patients enrolled in the intervention group compared to the control group, in episodes of respiratory rate alteration associated with noises > 45 dB (nursing diagnosis: risk of tachypnoea - RR >60 breaths per minute - correlated with environmental exposure to noises > 45dB).
Reduction of episodes of apnoea | Through study completion, an average of 2 year
  Reduction, in the patients enrolled in the intervention group compared to the control group, in episodes of apnoea associated with noises > 45 dB (nursing diagnosis: risk of apnoea - HR <100 bpm and SpO2 <90% - correlated with environmental exposure to noises > 45dB).

SECONDARY OUTCOMES:
Reduction in Language Development Alterations | From enrollment unitl 3 years of age
  The study will assess whether there is a reduction in language development issues in the intervention group compared to the control group. This evaluation will be conducted during a follow-up assessment at 3 years of age. The nursing diagnosis being considered is "risk of impaired verbal communication related to hospitalization in the NICU."
Reduction in Hearing Development Alterations | From enrollment unitl 3 months of age
  The study will also assess whether there is a reduction in hearing development issues in the intervention group compared to the control group. These evaluations will be conducted at a follow-up assessment at 3 months of age and any subsequent audiometric examinations. The nursing diagnosis being considered is "risk of compromised hearing development related to hospitalization in the NICU."

CONTACTS AND LOCATIONS:
Overall Officials: Simona Serveli, RN, Study Chair — Department of Health Profession, IRCCS Istituto Giannina Gaslini
Locations (1):
- IRCCS Istituto Giannina Gaslini, Genova, Genova, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data could be shared under a motivated request, only anonymised and grouped in databases.